CLINICAL TRIAL: NCT07095595
Title: The Effect of Education-based Patient Safety on Nursing Leaders' and Educators' Perceptions of Patient Safety Culture in Saudi Arabia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Ashwaq Talal Alahmadi, PhD student - Department of Nursing - Faculty of Medicine and Health Sciences, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALAHMADI-IRP-25-064
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Patient safety culture; safety culture; education; nursing

STUDY DESIGN:
Intervention Model Description: This a quasi-experimental with intervention or control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Interventional Group will receive a 5 day patient safety educational program
  Interventions: Other: Patient Safety Educational Program based on WHO Curriculum
- Control Group (No Intervention): Control group with no intervention

INTERVENTIONS:
Other: Patient Safety Educational Program based on WHO Curriculum — This study involves a structured 5-day educational program targeting nursing leaders and educators, with each day comprising 2 to 3 hours of instructional sessions. it will will include a combination of lectures, videos, group discussions, and case study analyses to enhance engagement and practical learning
  Arms: Interventional Group

SUMMARY:
This interventional study is aimed to examine the effect of an education-based patient safety on the perceptions of patient safety culture among nursing leaders and educators in one of the medical cities in Saudi Arabia. Participants will complete a perception survey before and three months after the educational program.

ELIGIBILITY:
Inclusion Criteria:

Nursing directors, deputy of nursing directors, head nurses, assistant head nurses, rotating shift nursing supervisors, nursing educators will be included in the current study.

Exclusion Criteria:

Bedside nurses were excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in Perceptions of Patient Safety Culture Among Nursing Leaders and Educators From Baseline to 3 Months Post-Intervention. | Baseline and 3 Months Post-Intervention
  This outcome measure will assess the change in nursing leaders' and educators' perceptions of patient safety culture before the educational intervention (baseline) and three months afterward. The assessment will be conducted using a validated patient safety culture survey instrument.

SECONDARY OUTCOMES:
Immediate Post-Intervention Feedback on Educational Program Effectiveness | Immediately Post-Intervention
  This outcome measure will assess participants' perceptions of the educational program's effectiveness immediately after completion. The questionnaire was developed and reviewed by WHO patient safety education team. Also, seven experts assessed the content validity using content validity index. The modifications were made in accordance with the suggestions provided by the jury.

CONTACTS AND LOCATIONS:
Locations (1):
- Medina Health Cluster, Madinah, Medina Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared, including participants' survey responses related to patient safety culture and program feedback. All personal identifiers (participants names, study city and name of institution) will not be shared.
  Based on IRP research team is not allowed to disclose personally identifiable data of the to any other party.